CLINICAL TRIAL: NCT04553952
Title: Evaluating the Distribution of Gingival Display and Possible Related Factors Resulting in Gummy Smile
Brief Title: The Distribution of Gingival Display and Possible Related Factors Resulting in Gummy Smile
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Mehtap Bilgin Çetin, DDS,PhD, Baskent University
Other Study IDs: MBilgin
Record Dates: First submitted 2020-09-07; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Gummy Smile

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gummy smile (GS(+))
  Interventions: Other: Measurement of gingival display
- Gumms smile(GS(-))
  Interventions: Other: Measurement of gingival display

INTERVENTIONS:
Other: Measurement of gingival display — All individuals were instructed to sit on a dental chair and the measurements were made by using a millimetric ruler. Next, the patients were grouped according to Liebart's classification by gingival display at maximum smile as follows:
  Class 1.Excessive gingival display (Gummy smile): ≥ 3mm gingival display Class 2.High smile line: 0-2 mm of gingival display Class 3. Average smile line: Dental papilla is visible. Class 4. Low smile line: Gingival margin, dental papilla is not visible at all.

SUMMARY:
This study primarily aimed to evaluate smile line distribution and prevalence of gummy smile in patients. The secondary purpose was to examine parameters that might be risk factors for gummy smile.

DETAILED DESCRIPTION:
this study primarily aimed to evaluate smile line distribution and prevalence of gummy smile in patients. The secondary purpose was to examine parameters that might be risk factors for gummy smile.Age, gender, marital status, medical history, and medication status of the patients were recorded. All individuals were instructed to sit on a dental chair and the measurments were made by using a millimetric ruler.Next, the patients were grouped according to Liebart's classification by gingival display at maximum smile as follows: Class 1.Excessive gingival display (Gummy smile): ≥ 3mm gingival display Class 2.High smile line: 0-2 mm of gingival display Class 3. Average smile line: Dental papilla is visible. Class 4. Low smile line: Gingival margin, dental papilla is not visible at all. Presence of altered passive eruption, short lip and hypermobile upper lip were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* presence of teeth in upper jaw
* Age between 18-65 years

Exclusion Criteria:

* Patients who have received and/or are receiving orthodontic treatment and patients who received gummy smile treatment were excluded.

Ages: 20 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who applied to Baskent University Faculty of Dentistry for seeking dental treatment
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2019-11-09 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
Measurement of gingival display | 1 minute
  All individuals were instructed to sit on a dental chair and the measurments were made by using a millimetric ruler. Next, the patients were grouped according to Liebart's classification by gingival display at maximum smile as follows:
  Class 1.Excessive gingival display (Gummy smile): ≥ 3mm gingival display Class 2.High smile line: 0-2 mm of gingival display Class 3. Average smile line: Dental papilla is visible. Class 4. Low smile line: Gingival margin, dental papilla is not visible at all.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University,Department of Dentistry, Ankara, Turkey (Türkiye)